CLINICAL TRIAL: NCT05438446
Title: Effect of Renal Denervation on Stress, Hypertension and Anxiety Management (ERSHAM Study) in Patients With Uncontrolled Hypertension
Brief Title: Effect of Renal Denervation on Stress, Hypertension and Anxiety Management
Acronym: ERSHAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Collaborators: ReCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor of Cardiology, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERSHAM
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Hypertension Arterial; Anxiety; Stress
MeSH Terms: conditions — Hypertension; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, interventional, 1:1 randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal Denervation Arm (Experimental): Endovascular ultrasound renal denervation (Paradise renal denervation system, ReCor, CA, USA) (RDN)
  Interventions: Procedure: Endovascular ultrasound renal denervation (Paradise renal denervation system, ReCor, CA, USA) (RDN)
- Control (No Intervention): The patient will not receive any interventional therapy

INTERVENTIONS:
Procedure: Endovascular ultrasound renal denervation (Paradise renal denervation system, ReCor, CA, USA) (RDN) — The ReCor Medical Paradise® Renal Denervation System (Paradise System) is CE-marked in countries accepting the CE mark, but Investigational in the USA.
  The system is a catheter-based device designed to use ultrasound energy to thermally ablate the afferent and efferent nerves surrounding the renal artery and serving the kidney.
  Arms: Renal Denervation Arm

SUMMARY:
The ERSHAM (Effect of Renal Denervation on Stress, Hypertension and Anxiety Management) is a single-center, interventional, open-label, randomized controlled trial that will be conducted at the Hypertension Unit "ESH Excellence Center'', 1st Cardiology Department of the Medical School of the National and Kapodistrian University of Athens at the General Hospital of Athens "Hippokration", which is the reference center for uncontrolled hypertension and for sympathetic renal denervation (RDN) in our region. Sixty (60) consecutive patients aged 30-70 years with uncontrolled arterial hypertension either under anti-hypertensive treatment with 1 drug [at least 50% of maximum manufacturer's recommended dosage of an angiotensin-converting enzyme inhibitor (ACEI)/ angiotensin II receptor blocker (ARB) or a calcium channel blocker (CCB)] or naïve from antihypertensive treatment and HADS (Hospital anxiety and depression scale) anxiety subscore ≥ 8 will be enrolled (Figure 1). Patients will be randomized in a 1: 1 ratio to endovascular ultrasound RDN (Paradise renal denervation system, ReCor, CA, USA) (RDN) (n= 30) or to control group (n= 30). Baseline clinical data, cardiovascular risk factors, medical history as well as medication will be recorded in each group. After the randomization, patients who will be randomized to RDN group will undergo a computed tomography angiography (CTA) or magnetic resonance angiography (MRA) of the renal arteries in order to assess whether the renal arteries' anatomy is suitable for RDN by using the Paradise system. The images of the CTA/MRA will be uploaded onto BIOCLINICA web-based portal in order to optimize device use (RDN catheter) and location of ablations. Patients will not change their antihypertensive medications during the 3 months follow -up. After that, their management will be evaluated based on the current 2018 ESC/ESH guidelines.

Possible RDN-related adverse events will be recorded during the follow-up period. Blood pressure (BP) will be measured by office BP measurements as well as 24-hour ambulatory blood pressure monitoring. Anxiety and depression will be evaluated by the self-assessment hospital anxiety and depression scale (HADS). Stress management will be evaluated via Perceived Stress Scale-14 (PSS-14). To assess the quality of life (QoL) the health status questionnaire (SF-12) will be used. The social readjustment rating scale will be used in order to evaluate the probability of developing a stress-related disorder during the follow-up period. Finally, a questionnaire for personal stress due to high blood pressure will be applied at the baseline and at the end of the follow-up period.

Patients will be followed-up for 6 months after the randomization. A total of three (3) follow-up visits for each patient will be scheduled during the 6-month follow-up period of the study [1st (adverse events review), 3rd, and 6th month after the randomization). If there is a failure in reaching the office BP <140/90mmHg at the 3rd and 6th month, the antihypertensive therapy will be reevaluated according to the current ESH/ESC Guidelines.

All patients will give written informed consent and the study will be organized according to ethical considerations, as described in the Declaration of Helsinki for human medical studies, and the protocol will be approved by the institutional medical ethics committee.

DETAILED DESCRIPTION:
Background

Uncontrolled hypertension (HTN) is of multifactorial origin and continues to represent a major public health issue. Sympathetic renal denervation (RDN) has been proposed as a promising, minimally invasive method to contribute to the improvement of HTN control. Data from recent multicenter randomized studies (SPYRAL HTN-OFF MED, SPYRAL HTN-ON MED, RADIANCE-HTN SOLO) provided solid data that RDN could achieve a clinically meaningful ambulatory and office blood pressure (BP) reduction in hypertensive patients with and without antihypertensive medications by using different technologies (radiofrequency energy or ultrasound energy to ablate the renal fibers). Beyond the BP control, RDN has demonstrated pleiotropic effects that occur partly independent of the observed BP reduction in various clinical settings (decreasing the "burden" of arrhythmias, decreasing left ventricular hypertrophy, increasing aortic compliance, improving sleep apnea and metabolic profile ), while recent data showed a positive impact in psychological disorders.

It is well known that the autonomic nervous system (ANS) plays a dominant role in both HTN and psychological disorders. In particular, dysfunction of the autonomic nervous system is considered to be the pathophysiological link between hypertension, depression, and anxiety. Sympathetic stimulation through mechanisms, such as, for example, renin secretion, is associated with elevated BP, while stressful life events are associated with depression and anxiety either contributing to or initiating the HTN. It is therefore perceived that the limitation of sympathetic activation could have a significant effect on both the control of the HTN and the management of psychological comorbidities leading to an improved quality of life (QoL).

Although the co-existence of increased sympathetic tone, HTN, and psychological disorders is well-established in the literature, the data concerning the effect of sympathetic RDN on stress management, anxiety disorders, and depression in patients with HTN is rather limited and is based mainly on case series and in non-randomized studies. In fact, the available data come from a study, which showed that RDN reduces anxiety disorders and depression, while it improves the quality of life in patients with resistant hypertension. However, a number of limitations accompanied the study: the patients had difficult-to-control hypertension (resistant or refractory hypertension), and most of the patients received antihypertensive drugs that can influence the patients' mood such as b-blockers.

Innovation

The investigators designed a randomized controlled trial [Effect of Renal Denervation on Stress, Hypertension and Anxiety Management (ERSHAM study)] in patients with uncontrolled hypertension, which aims to evaluate the effect of RDN on HTN, stress management, and anxiety disorders in patients with uncontrolled stage I HTN under no treatment or treatment with just one antihypertensive drug [angiotensin-converting enzyme inhibitor (ACEI)/ angiotensin II receptor blocker (ARB) or a calcium channel blocker (CCB)]. For this purpose, the investigators include patients with a baseline abnormal HADS score, while the investigators exclude patients under treatment with specific antihypertensive drugs that can affect aspects related to the quality of life such as diuretics and b-blockers.

Purpose

The purpose of this study is to test the hypothesis that renal sympathetic denervation has a short- (3 months) and long-term (6 months) positive effect on blood pressure lowering, stress management, and anxiety disorders and is associated with an improvement in quality of life in adult patients with uncontrolled arterial hypertension.

Design

Single-center, prospective, interventional, 1:1 randomized controlled trial

Medical device

The Paradise renal denervation system, Recor, CA, USA will be used in this clinical study. First in human evidence of the clinical safety and efficacy of the Paradise System was initially evaluated in the first-in-man REnal Denervation by Ultrasound transCatheter Emission (REDUCE) Trial, a single-center feasibility study initiated in 2011 and conducted at Vergelegen Medi-Clinic, South Africa. Subsequently, two multi-center, ReCor Medical Inc. sponsored post-market evaluations (the REALISE and ACHIEVE studies) were initiated in 2012, and 2013, respectively. An investigator-sponsored single-center study, RADIOSOUND-HTN, comparing radio frequency and ultrasound-based renal denervation utilizing the Paradise system was conducted in Germany between 2015 and 2018. In 2016, the RADIANCE HTN Study, a randomized, double-blind, two-cohort study evaluating the efficacy of the Paradise System in both primary hypertensive patients washed out of antihypertensive medications (SOLO Cohort)4 and resistant hypertensive patients (TRIO Cohort), was initiated. The RADIANCE-II pivotal study, a randomized, double-blind, single-cohort study in primary hypertensive patients washed out of antihypertensive medications was initiated in 2018.

The ERSHAM (Effect of Renal Denervation on Stress, Hypertension and Anxiety Management) is a single-center, interventional, open-label, randomized controlled trial that will be conducted at the Hypertension Unit "ESH Excellence Center'', 1st Cardiology Department of the Medical School of the National and Kapodistrian University of Athens at the General Hospital of Athens "Hippokration", which is the reference center for uncontrolled hypertension and for sympathetic renal denervation (RDN) in our region. Sixty (60) consecutive patients aged 30-70 years with uncontrolled arterial hypertension either under anti-hypertensive treatment with 1 drug (at least 50% of maximum manufacturer's recommended dosage of a ACEI/ARB or a CCB) or naïve from antihypertensive treatment and HADS (Hospital anxiety and depression scale) anxiety subscore ≥ 8 will be enrolled. Patients will be randomized in a 1: 1 ratio to endovascular ultrasound RDN (Paradise renal denervation system, ReCor, CA, USA) (RDN) (n= 30) or to control group (n= 30). Baseline clinical data, cardiovascular risk factors, medical history as well as medication will be recorded in each group. After the randomization, patients who will be randomized to RDN group will undergo a computed tomography angiography (CTA) or magnetic resonance angiography (MRA) of the renal arteries in order to assess whether the renal arteries' anatomy is suitable for RDN by using the Paradise system. The images of the CTA/MRA will be uploaded onto BIOCLINICA web-based portal in order to optimize device use (RDN catheter) and location of ablations. Patients will not change their antihypertensive medications during the 3 months follow -up. After that, their management will be evaluated based on the current 2018 ESC/ESH guidelines.

Possible RDN-related adverse events will be recorded during the follow-up period. Blood pressure (BP) will be measured by office BP measurements as well as ABPM. Anxiety and depression will be evaluated by the self-assessment hospital anxiety and depression scale (HADS). Stress management will be evaluated via the Perceived Stress Scale-14 (PSS-14), a 14-item scale that assesses the perception of stressful experiences by asking the respondent to rate the frequency of his/her feelings and thoughts related to events and situations that occurred over the previous month. To assess the quality of life (QoL) the health status questionnaire (SF-12) will be used. All the above psychometric scores are also validated in a Greek population. The social readjustment rating scale will be used in order to evaluate the probability of developing a stress-related disorder during the follow-up period. Finally, a questionnaire for personal stress due to high blood pressure will be applied at the baseline and at the end of the follow-up period.

Patients will be followed-up for 6 months after the randomization. A total of three (3) follow-up visits for each patient will be scheduled during the 6-month follow-up period of the study [1st month (adverse events review)], 3rd, and 6th month after the randomization]. If there is a failure in reaching the office BP <140/90mmHg at the 3rd and 6th month, the antihypertensive therapy will be reevaluated according to the current ESH/ESC Guidelines.

All patients will give written informed consent and the study will be organized according to ethical considerations, as described in the Declaration of Helsinki for human medical studies, and the protocol will be approved by the institutional medical ethics committee.

Blood Pressure Variability, Heart Rate Variability and Renal Denervation

BPV (Blood Pressure Variability) and HRV (Heart Rate Variability) are known to reflect the features of autonomic neural cardiovascular regulation, in particular the sympathetic and parasympathetic cardiac modulation and the so-called sympatho-vagal balance. BP (blood pressure) values change significantly over time as a result of the interaction between extrinsic environmental and behavioral factors and intrinsic cardiovascular regulatory mechanisms. Blood pressure variability (BPV) is a term describing the dynamic BP behavior over time, including both BP peaks and troughs. On the other hand, it is widely known that a sustained increase in BPV may also reflect alterations in cardiovascular regulatory mechanisms, often associated with pathological conditions, which are known to be associated with unfavorable hemodynamic, metabolic, cardiovascular, and renal effects, and to be responsible for cardiovascular complications.

The autonomic cardiovascular modulation (ACVM) is modified by renal denervation. The gold standard method to detect changes in ACVM is a battery of autonomic tests that investigate the integrity of the autonomic function by eliciting cardiac or vascular responses. These tests require the active participation of the subject and are not easy to be standardized. However, indexes of heart rate variability (HRV) can be easily obtained in controlled conditions without the patients' active participation. Since different HRV measures reflect the functioning of the autonomic nervous system, there is a rising interest in using HRV indexes to quantify the changes in ACVM induced by RDN.

Despite the fact that RDN studies have different types of BP measurement available (including ambulatory BP monitoring, ABPM, and home BP monitoring, HBPM) both at baseline and at different times after the procedure, it is still unknown whether individuals with increased BPV at baseline (after accounting for their mean BP levels) or/and with increased HRV at baseline (after accounting for their mean HR levels) are those better responders to RDN, in term of BP reduction and reduction of BPV/HRV.

Obstructive Sleep Apnea and Renal Denervation

Patients with obstructive sleep apnea (OSA) present high levels of psychological stress and anxiety and depressive symptoms. OSA is a common comorbidity in patients with arterial hypertension (HTN), especially in patients with resistant HTN9. OSA is linked to sympathetic nervous system activation, and patients with OSA frequently have elevated blood pressure (BP), increased BP variability, and nocturnal BP surges. Recent evidence associates sympathetic tone with the severity of hypertension and OSA.

Renal sympathetic denervation (RDN), by decreasing sympathetic tone, has the potential to decrease OSA severity. More importantly, OSA patients appeared to be more responsive to RDN. In a posthoc analysis of SIMPLICITY-HTN 3 trial, RDN patients had lower 6-month office systolic BP than sham control patients (-17.0±22.4 vs. -6.3±26.1 mmHg, P=0.01) but not in patients without OSA (-14.7±24.5 vs. -13.4±26.4 mmHg, P=0.64), P=0.07 for the interaction between treatment arm and OSA status.

On the other hand, RDN seems to improve OSA severity, and showed, for the first time, that catheter-based renal sympathetic denervation lowers BP in resistant hypertensive patients with OSA. They speculated that reduced sodium and water retention may result in less edema of the upper airway, with diminished upper airway resistance and mitigation of airway collapse. Alternatively, they considered the possibility that the fall in BP may itself contribute to the attenuation of sleep apnea. This may be mediated by baroreflex deactivation inducing changes in chemoreflex modulation of breathing control or by direct effects of lower BP on central ventilator or airway control mechanisms.

However, the evidence for the positive effects of RDN in OSA patients is limited and it is based mainly on small observational studies that assessed this hypothesis. In addition, the precise mechanisms underlying the association between RDN and improvement in OSA severity are unclear, although these potential mechanisms certainly raise suspicion of association.

In addition to the ERSHAM protocol, all the enrolled patients will undergo 24h ABPM, 24h holter ECG, and noninvasively BP/HR measures with FINAPRES system by obtaining recordings during a 15-minute period of supine rest (SUP) followed by 10 minutes of standing, at baseline and at three months after RDN. In parallel to that, the investigators will obtain additional indexes of HRV through 24h holter ECG recordings and indexes of BPV through 24h ABPM recordings obtained before and three months after the procedure, in order to investigate whether those with altered BPV/HRV at baseline indicating an increased sympatho-vagal balance are those better responding in term of BP reduction and normalization of sympathovagal on BPV and HRV to RDN. All patients will be offered a cuffless BP monitoring device (Aktiia) to obtain a weekly BP monitoring at baseline and at 3 months after RDN". Day-to-day BPV will be evaluated.

Moreover, all the enrolled patients will undergo a full-night polysomnography using the SOMNOscreenTM device during unattended home Polygraphy at baseline and 3 months after randomization. The device continuously monitors a) Airflow with Nasal Cannula, or CPAP mask pressure; b) Thoracic/Abdominal Effort using two strain gauges; c) Snoring via nasal Cannula; d) Oxygen Saturation; e) Pulse Rate (pulse oximetry); f) Body Position, via a sensor in the cable box.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 30-70 years with arterial hypertension diagnosed at least 3 months prior to the inclusion.
* Office blood pressure (OBP) >140/90mmHg and <160/100 mmHg
* Either no baseline hypertension treatment or hypertension treatment with one drug. The antihypertensive treatment will include a renin-angiotensin system (RAS) blocker [either an angiotensin-converting enzyme inhibitor (ACEI) or an angiotensin receptor blocker (ARB)] or a calcium channel blocker (CCB).
* Unchanged antihypertensive therapy during the prior 8 weeks.
* Patients with baseline anxiety subscore ≥ 8 according to the Hospital Anxiety and Depression Scale (HADS)

Exclusion Criteria:

* Patients with secondary arterial hypertension or under treatment with b-blockers, diuretics, mineralocorticoid receptors antagonists (MRAs) or a centrally acting alpha-adrenergic agonist.
* Patients under treatment with antidepressants and/or anxiolytic drugs.
* Patients with a glomerular filtration rate (eGFR)] <45 ml / min / 1.73 m2 calculated using the CKD-EPI formula15.
* Patients with evidence of any of the following criteria on either renal artery side:

  * Main renal artery diameter < 3.0 mm or > 8 mm
  * Main renal treatable artery length < 20 mm
  * Presence of renal artery stenosis of any origin ≥ 30%
  * Accessory arteries with diameter ≥ 2mm <3.0 mm
  * Calcification in renal arteries at location where energy is to be delivered
  * A single functioning kidney
  * Prior renal denervation procedure
  * Presence of abnormal kidney tumors
  * Renal artery with aneurysm
  * Pre-existing renal stent or history of renal artery angioplasty
  * Pre-existing aortic stent or history of aortic aneurysm
  * Fibromuscular disease of the renal arteries
  * Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter
* Patients with a history of acute coronary syndrome or stroke during the previous six months or Scheduled coronary interventional therapy during the next six months.
* Patients with permanent atrial fibrillation, chronic heart failure and NYHA functional status II-IV, Cancer under therapy (radiotherapy, chemotherapy, immunotherapy)
* Patients with life expectancy <1 year (at the time of inclusion).
* Pregnant women or women who are planning to become pregnant.
* Patients who do not provide written consent to participate in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety 1 | From baseline (Screening Visit -1) at 3 months (Visit 2) of the follow-up period.
  Change in the Hospital Anxiety and Depression Scale (HADS) anxiety subscore
Hypertension | From baseline (Visit 0) at 3 months (Visit 2) of the follow-up period.
  Change in the 24h systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Anxiety 2 | From baseline (Screening Visit -1) at 6 months (Visit 3) of the follow-up period.
  Change in the Hospital Anxiety and Depression Scale (HADS) anxiety subscore
Depression | From baseline (Screening Visit -1) at 3 (Visit 2) and 6 months (Visit 3) of the follow-up period
  Change in the Hospital Anxiety and Depression Scale (HADS) depression subscore
Stress | From baseline (Visit 0) at 3 (Visit 2) and 6 months (Visit 3) of the follow-up period.
  Change in the Perceived Stress Scale-14 (PSS-14)
Physical and Mental Health | From baseline (Visit 0) at 3 (Visit 2) and 6 months (Visit 3) of the follow-up period.
  Change in the Short Form 12 Health Survey (SF-12) scale
Office Blood Pressure 1 | From baseline (Visit 0) at 3 months (Visit 2) of the follow-up period.
  Change in the office systolic and diastolic blood pressure
Office Blood Pressure 2 | From baseline (Visit 0) at 6 months (Visit 3) of the follow-up period.
  Change in the office systolic and diastolic blood pressure
Ambulatory Blood Pressure Monitoring (ABPM) | From baseline (Visit 0) at 6 months (Visit 3).
  Change in the 24h systolic and diastolic blood pressure
Heart Rate | From baseline (Visit 0) at 3 (Visit 2) and 6 months (Visit 3) of the follow-up period.
  Change in the patients' heart rate
Blood Pressure Variability (BPV) | From baseline (Screening Visit -1) at 3 months (Visit 2) of the follow-up period
  Change in the BPV
Heart Rate Variability (HRV) | From baseline (Screening Visit -1) at 3 months (Visit 2) of the follow-up period
  Change in the HRV
Apnea- Hypopnea | From baseline (Screening Visit -1) at 3 months (Visit 2) of the follow-up period.
  Change in the Apnea- Hypopnea Index

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tsioufis, MD, PhD, Principal Investigator — Hippokration Hospital, Athens, Greece
Locations (1):
- Hippokration Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsioufis C, Ziakas A, Dimitriadis K, Davlouros P, Marketou M, Kasiakogias A, Thomopoulos C, Petroglou D, Tsiachris D, Doumas M, Skalidis E, Karvounis C, Alexopoulos D, Vardas P, Kallikazaros I, Stefanadis C, Papademetriou V, Tousoulis D. Blood pressure response to catheter-based renal sympathetic denervation in severe resistant hypertension: data from the Greek Renal Denervation Registry. Clin Res Cardiol. 2017 May;106(5):322-330. doi: 10.1007/s00392-016-1056-z. Epub 2016 Dec 12. PMID 27957627
- [Background] Schmieder RE, Mahfoud F, Azizi M, Pathak A, Dimitriadis K, Kroon AA, Ott C, Scalise F, Mancia G, Tsioufis C; Members of the ESH Working Group on Interventional Treatment of Hypertension. European Society of Hypertension position paper on renal denervation 2018. J Hypertens. 2018 Oct;36(10):2042-2048. doi: 10.1097/HJH.0000000000001858. PMID 30015759
- [Background] Papademetriou V, Doumas M, Tsioufis K. Renal Sympathetic Denervation for the Treatment of Difficult-to-Control or Resistant Hypertension. Int J Hypertens. 2011;2011:196518. doi: 10.4061/2011/196518. Epub 2011 Mar 30. PMID 21629864
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590
- [Background] Lenski D, Kindermann I, Lenski M, Ukena C, Bunz M, Mahfoud F, Bohm M. Anxiety, depression, quality of life and stress in patients with resistant hypertension before and after catheter-based renal sympathetic denervation. EuroIntervention. 2013 Oct;9(6):700-8. doi: 10.4244/EIJV9I6A114. PMID 24169132
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Venkataraman S, Vungarala S, Covassin N, Somers VK. Sleep Apnea, Hypertension and the Sympathetic Nervous System in the Adult Population. J Clin Med. 2020 Feb 21;9(2):591. doi: 10.3390/jcm9020591. PMID 32098169
- [Background] Parati G, Ochoa JE, Lombardi C, Bilo G. Assessment and management of blood-pressure variability. Nat Rev Cardiol. 2013 Mar;10(3):143-55. doi: 10.1038/nrcardio.2013.1. Epub 2013 Feb 12. PMID 23399972
- [Background] Seravalle G, D'Arrigo G, Tripepi G, Mallamaci F, Brambilla G, Mancia G, Grassi G, Zoccali C. Sympathetic nerve traffic and blood pressure changes after bilateral renal denervation in resistant hypertension: a time-integrated analysis. Nephrol Dial Transplant. 2017 Aug 1;32(8):1351-1356. doi: 10.1093/ndt/gfx200. PMID 28810724
- [Background] Michopoulos I, Douzenis A, Kalkavoura C, Christodoulou C, Michalopoulou P, Kalemi G, Fineti K, Patapis P, Protopapas K, Lykouras L. Hospital Anxiety and Depression Scale (HADS): validation in a Greek general hospital sample. Ann Gen Psychiatry. 2008 Mar 6;7:4. doi: 10.1186/1744-859X-7-4. PMID 18325093